CLINICAL TRIAL: NCT03874585
Title: Text Messaging-Based Smoking Cessation Program for Homeless Youth
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Principal Investigator, Joan Tucker, Senior Behavioral Scientist, RAND
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27IP-0051
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Condition (Active Comparator): Participants in the standard condition will receive a 30-minute group-based smoking cessation counseling session based on the 5 A's approach (Ask; Advise; Assess; Assist; Arrange) and free nicotine replacement.
  Interventions: Behavioral: Group counseling and nicotine replacement
- Enhanced Condition (Experimental): Participants in the standard condition will receive a 30-minute group-based smoking cessation counseling session based on the 5 A's approach (Ask; Advise; Assess; Assist; Arrange), free nicotine replacement, and the 6-week text messaging intervention.
  Interventions: Behavioral: Group counseling, nicotine replacement, and text messaging support

INTERVENTIONS:
Behavioral: Group counseling and nicotine replacement — Participants will receive a 30-minute group smoking cessation counseling session and a supply of nicotine replacement.
  Arms: Standard Condition
Behavioral: Group counseling, nicotine replacement, and text messaging support — Participants will receive a 30-minute group smoking cessation counseling session, a supply of nicotine replacement, and the 6-week text messaging intervention to provide ongoing support for quitting
  Arms: Enhanced Condition

SUMMARY:
Unaccompanied homeless youth smoke at much higher rates than non-homeless adolescents and young adults. Many homeless youth smokers are motivated to quit; yet, strategies specifically developed for this vulnerable population are lacking. This study will develop and pilot test a text messaging intervention (also known as a TMI) to help homeless youth quit smoking. Text messaging can provide ongoing support for homeless youth during a quit attempt, which is important given that these youth tend to be highly mobile and lack regular access to health services. Participants in this study will be homeless youth who currently smoke and are motivated to quit smoking. All participants will receive a 30-minute group-based smoking cessation counseling session and a nicotine replacement product. Half of these smokers will also receive the TMI, for 6 weeks following the group counseling session, which will provide ongoing support for quitting. The main goal of this study is to investigate whether receiving the TMI results in greater reductions in cigarette smoking over a 3-month period compared to receiving the group counseling session alone.

ELIGIBILITY:
Inclusion Criteria:

* between ages of 18-25
* seeking services at one of the participating drop-in centers for homeless youth
* smoked at least 5 cigarettes per day on at least 20 days in the past month
* motivated to quit in next 30 days
* has a cell phone to receive text messages and willing to receive text messages

Exclusion Criteria:

* currently pregnant or breastfeeding, or planning to become pregnant or breastfeed in the next 6 months
* has a medical condition (based on self-report) which would prevent using the nicotine replacement product
* used pharmacotherapy to reduce or stop smoking in the past 30 days
* currently receiving other smoking cessation services

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-05-21 (Actual)

PRIMARY OUTCOMES:
90 day continuous abstinence | 90 days
  Participants will self-report whether they have smoked any cigarettes between baseline and 3-month follow-up
7 day abstinence | 7 days
  Participants will self-report whether they have smoked any cigarettes in the past 7 days. Self-reported abstinence will be biochemically verified.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - My Friend's Place, Los Angeles, California
  - Los Angeles LGBT Center Youth Center, Los Angeles, California
  - Safe Place for Youth, Venice, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pedersen ER, Linnemayr S, Shadel WG, Zutshi R, DeYoreo M, Cabreros I, Tucker JS. Substance Use and Mental Health Outcomes from a Text Messaging-Based Intervention for Smoking Cessation Among Young People Experiencing Homelessness. Nicotine Tob Res. 2022 Jan 1;24(1):130-134. doi: 10.1093/ntr/ntab160. PMID 34375409
- [Derived] Tucker JS, Linnemayr S, Pedersen ER, Shadel WG, Zutshi R, DeYoreo M, Cabreros I. Pilot Randomized Clinical Trial of a Text Messaging-Based Intervention for Smoking Cessation Among Young People Experiencing Homelessness. Nicotine Tob Res. 2021 Aug 29;23(10):1691-1698. doi: 10.1093/ntr/ntab055. PMID 33852730
- [Derived] Linnemayr S, Zutshi R, Shadel W, Pedersen E, DeYoreo M, Tucker J. Text Messaging Intervention for Young Smokers Experiencing Homelessness: Lessons Learned From a Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Apr 1;9(4):e23989. doi: 10.2196/23989. PMID 33792551
- [Derived] Tucker JS, Pedersen ER, Linnemayr S, Shadel WG, DeYoreo M, Zutshi R. A text message intervention for quitting cigarette smoking among young adults experiencing homelessness: study protocol for a pilot randomized controlled trial. Addict Sci Clin Pract. 2020 Feb 19;15(1):11. doi: 10.1186/s13722-020-00187-6. PMID 32075695